CLINICAL TRIAL: NCT04474340
Title: COVID-19 Convalescent Plasma Treatment in SARS-CoV-2 Infected Patients: Multicenter Interventional Study
Brief Title: COVID-19 Convalescent Plasma Treatment in SARS-CoV-2 Infected Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Health, Kuwait (Other Government)
Responsible Party: Principal Investigator, Sondus AlSharidah, Sondus Alsharidah, Ministry of Health, Kuwait
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOHKuwait
Record Dates: First submitted 2020-07-15; First posted 2020-07-16 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Moderate COVID-19 Pneumonia, Severe COVID-19 Pneumonia; Pneumonia, Viral
Keywords: convalescent plasma; respiratory infection; COVID-19; SARS-CoV-2; pneumonia
MeSH Terms: conditions — Pneumonia, Viral; Respiratory Tract Infections; COVID-19; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCP patients (Experimental): 1. Patient has to fulfil the inclusion/exclusion criteria of the ward or the ICU
  2. Valid consent.
  3. Request the CCP from the central blood bank (200-250 ml/dose - can be repeated again in 12 hours) this is through the local hospital blood bank.
  How to transfuse CCP:
  1. Dose required is 200-250 ml/hr (one dose, can be repeated in 12 hrs), max total 500ml.
  2. Premedication prior to administration of CCP (Acetaminophen, diphenhydramine,steriods) or according to hospital guidelines.
  Interventions: Drug: COVID-19 Convalscent Plasma
- Control (No Intervention): Standard COVID-19 treatment.

INTERVENTIONS:
Drug: COVID-19 Convalscent Plasma — The source convalescent plasma is typically collected from individuals who have recovered from COVID-19 which contains antibodies titer against SARS-CoV-2 and is administered to patients with COVID-19. Donor eligibility criteria and qualification are based on American Accredited Blood Banks ( AABB) standards , including questionnaires and relevant transfusion-transmitted infections testing are performed. Furthermore, pathogen inactivation will be performed for each unit, CCP was only collected from individuals who meet all donor eligibility requirements (21 CFR 630.10 and 21 CFR 630.15). Donors must be found positive at a diagnostic test of nasopharyngeal swab at the time of illness and positive serological test for SARS-CoV-2 antibodies after recovery. All donors should have negative HLA antibodies.
  Arms: CCP patients

SUMMARY:
Due to the limitations of COVID-19 treatment and in the absence of licensed antiviral for COVID-19, the historical choice of therapeutic convalescent plasma (CP) is considered especially against RNA viruses .It was known that convalescent plasma does not only neutralize the pathogens but provide passive immunomodulatory properties that allows the recipient to control the exaggerated inflammatory cascade. However, still there is a lack of understanding of the mechanism of action of CCP therapeutic components. Reports from open label trials and case series show that CCP is safe and might be effective in severe cases with COVID-19 . Therefore, the World health organisation (WHO) and Food and Drug Administration (FDA) issued guidelines for the CCP usage and standardised the donor selection , which was further supported by Emergency use Authorisation (EUA) .

Therefore, the aim in the current study is to assess the effect of CCP on time to clinical improvement, hospital mortality and to evaluate the changes on oxygen saturation and laboratory markers (lymphocyte counts and C-reactive protein) compared with standard treatment alone in patients with moderate or severe COVID-19 disease.

DETAILED DESCRIPTION:
This is a prospective multicenter interventional observational study will be conducted in 4 major tertiary hospitals (Al-Sabah, Farwaniya , Mubarak Al-Kabeer and Jahra) in Kuwait .

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years old ( those who are younger are involved after case based discussion)
2. Confirmed laboratory diagnosis with SARS-CoV-2 ,and admission diagnosis of SARS-CoV-2.
3. Patients with moderate or severe COVID-19 (moderate COVID-19 disease defined as the presence of any signs of pneumonia (fever, cough, dyspnoea fast breathing) including SpO2 >90 on room air , but no signs of severe pneumonia (severe pneumonia have the above plus one of the following: respiratory rates >30 breaths/minutes or SpO2<90% on room air), or admission to intensive care unit (ICU) for respiratory support (i.e.high flow nasal cannula, non-invasive mechanical ventilation and intubation).

Exclusion Criteria:

1. -Contraindication to transfusion (volume overload, history of anaphylaxis to blood products).
2. - Patients presenting with acute severe multiorgan failure, hemodynamic instability.

3- Severe disseminated coagulopathy (DIC), septic shock and those with expected survival of less than 48 hours.

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-05-21 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to clinical improvement | 30 days
  Time to clinical improvement is defined as a time frame from CCP administration till 30 days or discharge, defined as a 2-grade decrease on an ordinal WHO clinical scale . The WHO clinical scale based on the following 7-grade ordinal levels: 1= ambulatory, independent; 2= ambulatory with assistance; 3=hospitalised, not requiring supplemental oxygen; 4= hospitalised, requiring supplemental oxygen; 5= hospitalised, requiring nasal high-flow oxygen therapy, noninvasive mechanical ventilation, or both; 6= hospitalised, requiring extracorporeal membrane oxygenation, invasive mechanical ventilation, or both; and 7= death.

SECONDARY OUTCOMES:
All cause mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Sondus AlSharidah, MD, Principal Investigator — MOH
Locations (1):
- Ministry Of Health, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol